CLINICAL TRIAL: NCT06241014
Title: Effects of Mulligan Mobilization With and Without Sling Exercises on Pain and Disability in Non-specific Neck Pain
Brief Title: Effects of Mulligan Mobilization With and Without Sling Exercises in Non-specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0157
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain
Keywords: Mulligan Exercises; Sling Exercises; Neck disability
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Group A will be treated with mulligan mobilizations and Sling exercises. (Experimental): Group A: In this group, Subjects will be treated with Mulligan mobilizations along with sling exercises. Mulligan mobilizations include SNAGs. Participants will receive 3 sets of mulligan mobilization techniques per session, each set involving 10 times repetition of the exercise. The interval between the sets will be 15 to 20 seconds. The technique will be repeated total of six times, having two sessions per week for 3 weeks. The sling exercise program will also be applied for 3 weeks, 2 times a week for 20 minutes per day.
  Interventions: Other: Mulligan Mobilization and Sling Exercises
- Group B: Group B will be treated with mulligan mobilizations alone. (Active Comparator): Group B: In this group, Subjects will be treated with Mulligan mobilizations and sling exercises. Mulligan mobilizations include SNAGs. Participants will receive 3 sets of mulligan mobilization techniques per session, each set involving 10 times repetition of the exercise. The interval between the sets will be 15 to 20 seconds. The technique will be repeated a total of six times, having two sessions per week for 3 weeks.
  Interventions: Other: Mulligan Mobilization

INTERVENTIONS:
Other: Mulligan Mobilization and Sling Exercises — Mulligan mobilizations along with sling exercises. Mulligan mobilizations include SNAGs. Participants will receive 3 sets of mulligan mobilization techniques per session, each set involving 10 times repetition of the exercise. The interval between the sets will be 15 to 20 seconds. The technique will be repeated total of six times having two sessions per week for 3 weeks. For the sling exercise, the sling exercise program will also be applied for 3 weeks, 2 times a week for 20 minutes per day. To perform the exercise, the subjects will be instructed with a demonstration and explanation.
  Arms: Group A: Group A will be treated with mulligan mobilizations and Sling exercises.
Other: Mulligan Mobilization — Mulligan Mobilization
  Arms: Group B: Group B will be treated with mulligan mobilizations alone.

SUMMARY:
Neck pain is one of the common musculoskeletal problems. People with neck pain can have difficulties with daily activities and be limited in work and social participation. Main symptoms of people with neck pain include pain, decreased range of motion (ROM), muscle weakness and dysfunction. Common neck pain causes include degenerative disc disease, herniated disc disease, cervical radiculopathies, myofascial pain syndrome and viral infections. Muscular strains, postural and ergonomics are also related to neck pain and whiplash injuries. The onset of pain may be insidious or may follow trauma, and it may be recurrent or persistent in nature. Ideally, the pain goes away in 1-3 weeks, but in some cases it persists and become chronic neck pain. The aim of this study is to compare the effects of mulligan mobilization with and without sling exercises on pain, and disability in non-specific neck pain. Non-specific neck pain reduces range of motion which may be linked to mechanical restriction between two or more vertebrae and muscular spasm.

DETAILED DESCRIPTION:
Participants who will meet the inclusion criteria will be recruited by convenience sampling technique and will be allocated to groups by simple randomization process by sealed opaque enveloped labeled as 1 for Group A and 2 for Group B.

After taking consent from the participants with non-specific neck pain of both genders will be randomized into two equal groups. Subjects from physical therapy department will be assessed with neck disability index, goniometer and Numeric pain rating scale. At start of study, a formal educational session, lasting about 30 min will be given by physiotherapist.

Group A: In this group, Subjects will be treated with Mulligan mobilizations along with sling exercises. Mulligan mobilizations include SNAGs. Participants will receive 3 sets of mulligan mobilization techniques per session, each set involving 10 times repetition of the exercise. The interval between the sets will be 15 to 20 seconds. The technique will be repeated total of six times having two sessions per week for 3 weeks.

For the sling exercise, the sling exercise program will also be applied for 3 weeks, 2 times a week for 20 minutes per day. To perform the exercise, the subjects will be instructed with a demonstration and explanation. In supine position, the head will be supported by an inelastic sling and the therapist will hold the cervical vertebral portion softly with two hands. Therapist will pull the cervical vertebral portion and back of the head softly. The subjects will maintain this for 6-7 seconds and relax slowly. In the second technique, Subjects will be positioned in supine lying position with the cervical spine in a neutral position on the sling device. One hand of the therapist contacts and fixes the transverse process of C1 (both), while the other hand grabs the occiput and applies mobilization in the dorsal direction. Subjects in this group will be applied with passive mobilization for 3 min to the segment (occiput-C1). In the same posture the subjects will be instructed to perform a flexion motion at (occiput-C1). The therapist will guide the optimal segmental movement through the hand. This intervention will also be performed 3 times for 1 min, with an interval of 1 min. Similarly, In prone position the forehead will be placed on an inelastic sling. The therapist will hold the cervical vertebral portion with two hands softly. The therapist will pull the cervical vertebral portion toward the upper direction at the same time. The patient will maintain this for 6-7 seconds and relax slowly. Each movement will be repeated 10 times

ELIGIBILITY:
Inclusion Criteria:

* Age between 25-50 years.
* Having neck pain for at least 2 weeks
* Pain intensity of at least 2 on NPRS
* Greater than or equal to 15 points on the neck disability index (NDI)
* Having primary complaint of non-specific neck pain

Exclusion Criteria:

* History of Cervical surgery
* Cervicogenic headache
* Previous cervical spine surgery
* Serious Spinal pathology (like tumor, infection, and dislocation)
* Traumatic injuries (e.g., contusion, fracture, and whiplash injury)
* Vascular diseases and Neurologic disorders (e.g., trigeminal neuralgia)
* Concomitant medical diagnosis of any primary headache (vertigo, VBI or migraine)
* And clinical diagnosis of cervical radiculopathy, Spinal stenosis or myelopathy.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | upto 4 weeks
  Patient level of pain will be assessed using this scale. In a Numerical Rating Scale (NRS), this scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain" patients are asked to circle the number between 0 and 10, that fits best to their pain intensity.
  NRS scores ≤ 5 correspond to mild, scores of 6-7 to moderate and scores ≥8 to severe pain in terms of pain-related interference with functioning.
Neck Disability Index | upto 4 weeks
  NDI is a simple ten-item questionnaire used to assess patients with neck pain. The questionnaire was devised and validated in English. It consists of ten questions each with six answers (scoring 0-5 points). The NDI has a fair to moderate test-retest reliability in patients with mechanical neck pain.
Universal Goniometer | upto 4 weeks
  A goniometer will be used in the study to measure shoulder flexion, internal rotation and external rotation.
  Goniometer is an instrument that measures the available range of motion at a joint. To .measure the range of motion physical therapists most commonly use a goniometer. Therapist can use a goniometer to assess what the range of motion is at the initial assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Abu Zar, MS, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Pro Care Health Clinic, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buyukturan O, Buyukturan B, Sas S, Kararti C, Ceylan I. The Effect of Mulligan Mobilization Technique in Older Adults with Neck Pain: A Randomized Controlled, Double-Blind Study. Pain Res Manag. 2018 May 15;2018:2856375. doi: 10.1155/2018/2856375. eCollection 2018. PMID 29861800
- [Background] Kim SY, An CM, Cha YS, Kim DH. Effects of sling-based manual therapy on cervicothoracic junction in patients with neck pain and forward head posture: A randomized clinical trial. J Bodyw Mov Ther. 2021 Jul;27:447-454. doi: 10.1016/j.jbmt.2021.03.007. Epub 2021 Mar 19. PMID 34391270
- [Background] Lin KY, Tsai YJ, Hsu PY, Tsai CS, Kuo YL. Effects of Sling Exercise for Neck Pain: A Systematic Review and Meta-Analysis. Phys Ther. 2021 Aug 1;101(8):pzab120. doi: 10.1093/ptj/pzab120. PMID 33929540
- [Background] Lee J-D, Shin W-S. Immediate effects of neuromuscular control exercise on neck pain, range of motion, and proprioception in persons with neck pain. Physical Therapy Rehabilitation Science. 2020;9(1):1-9.
- [Background] Manzoor A, Anwar N, Khalid K, Haider R, Saghir M, Javed MA. Comparison of effectiveness of muscle energy technique with Mulligan mobilization in patients with non-specific neck pain. J Pak Med Assoc. 2021 Jun;71(6):1532-1524. doi: 10.47391/JPMA.981. PMID 34111066
- [Background] He Y, Sun W, Zhao X, Ma M, Zheng Z, Xu L. Effects of core stability exercise for patients with neck pain: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2019 Nov;98(46):e17240. doi: 10.1097/MD.0000000000017240. PMID 31725601
- [Background] Kim YW, Kim NY, Chang WH, Lee SC. Comparison of the Therapeutic Effects of a Sling Exercise and a Traditional Stabilizing Exercise for Clinical Lumbar Spinal Instability. J Sport Rehabil. 2018 Jan 1;27(1):47-54. doi: 10.1123/jsr.2016-0083. Epub 2018 Jan 17. PMID 27992296
- [Background] Mun D-J, Oh H-J, Lee S-H. Effects of sling exercise on pain, trunk strength, and balance in patients with chronic low back pain. The Journal of Korean Physical Therapy. 2022;34(3):110-5.